CLINICAL TRIAL: NCT05621408
Title: Attention Training Technique in Treatment of Anxiety and Depression in Coronary Heart Disease Patients -a Randomized Controlled Trial With 6 Months Follow-up
Brief Title: Attention Training Technique in Treatment of Anxiety and Depression in Coronary Heart Disease Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: Oslo University Hospital (Other); University of Oslo (Other); The Hospital of Vestfold (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 52002
Record Dates: First submitted 2022-11-02; First posted 2022-11-18 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Depression, Anxiety; Coronary Artery Disease
MeSH Terms: conditions — Depression; Anxiety Disorders; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attention Training Techniqe (Experimental): The treatment manual will consist of up to six weekly group sessions with 45-90 minutes duration.
  Interventions: Behavioral: Attention Training Technique
- Wait-list control (No Intervention): The wait-list control condition will not receive any psychological intervention during the six weeks waiting period. Subsequently, this group will also receive the intervention if the study entry criteria is still fulfilled

INTERVENTIONS:
Behavioral: Attention Training Technique — Attention Training Technique is a six weeks psychological intervention provided by trained professionals
  Arms: Attention Training Techniqe

SUMMARY:
Anxiety and depression are associated with work disability, lower participation rate in cardiac rehabilitation and unfavourable life style changes following a coronary heart disease (CHD) event. The prevalence of clinically significant symptoms of depression and anxiety in CHD patients has been estimated to 30-50%. Furthermore, depression and anxiety are associated with a significant increased risk of subsequent major adverse cardiovascular events and mortality in CHD patients. Psychological interventions for anxiety and depression in CHD patients have demonstrated small and uncertain effects of symptoms, and no effect on cardiovascular outcomes. Therefore, testing the effectiveness of specific psychological interventions that may affect central mechanisms for cardiovascular outcomes, has been requested. The Attention training (ATT) Study is a randomized controlled trial comparing group-attention training to wait-list control in 64 patients who experience significant anxiety and depression after a CHD event. It will also be explored whether reduction in psychological symptoms is correlated with changes in biological markers with a potential link to cardiovascular outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Established coronary heart disease as main somatic disease
* >=8 on either HADS-anxiety or depression subscale
* Age 18 - 65 years
* The ability to understand and speak Norwegian language,
* Willingness and ability to give informed consent.

Exclusion Criteria:

* Current or past neurological illness
* Traumatic brain injury
* Current alcohol and/or substance dependency disorders
* Psychotic disorders
* Bipolar disorders
* Developmental disorders
* Mental retardation
* Cognitive impairment which precludes informed consent/ability to participate
* Acute suicidality
* Life-expectancy less than 12 months
* Concurrent psychological intervention for emotional distress
* Antidepressant or anxiolytic medication initiated during previous 8 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Changes in Hospital Anxiety and Depression -anxiety subscale score and Hospital Anxiety and Depression -depression subscale score | Up to six weeks and six months after randomization
  Changes in Hospital Anxiety and Depression -anxiety subscale score and Hospital Anxiety and Depression -depression subscale scores within and between the two treatment arms. Scores range 0-21, higher scores indicate more symptoms
Differences in proportion with Hospital Anxiety and Depression -anxiety and Hospital Anxiety and Depression-depression subscale scores <8 | Up to six weeks and six months after randomization
  Differences in proportion with Hospital Anxiety and Depression -anxiety subscale and Hospital Anxiety and Depression -depression subscale scores <8 within and between the two treatment arms. Scores >=8 indicate signicant symptoms

SECONDARY OUTCOMES:
Changes in rumination scores | Up to six weeks and six months after randomization
  Changes in rumination scores assessed by the Ruminative Response scale within and between the two treatment arms. Scores range from 22-88, higher scores indicate more symptoms
Changes in worry scores | Up to six weeks and six months after randomization
  Changes in worry scores assessed by the Penn State Worry Questionnaire within and between the two treatment arms. Scores range 16-80, higher scores indicate more symptoms
Changes in Positive Beliefs about Rumination Scale scores | Up to six weeks and six months after randomization
  Changes in Positive Beliefs about Rumination scores assessed by the Positive Beliefs about Rumination Questionnaire within and between the two treatment arms. Scores range 9-36, higher scores indicate stronger beliefs
Changes in Negative Beliefs about Rumination Scale scores | Up to six weeks and six months after randomization
  Changes in Negative Beliefs about Rumination scores assessed by the Negative Beliefs about Rumination Questionnaire within and between the two treatment arms. Scores range 13-52, higher scores indicate stronger beliefs
Changes in Metacognitions Questionnaire-30 scores | Up to six weeks and six months after randomization
  Changes in Metacognitions assessed by the Metacognitions Questionnaire-30 within and between the two treatment arms. Scores range 0-21, higher scores indicate more symptoms . Scores range 30-120, higher scores indicate stronger beliefs
Changes in type d personality and its traits negative affectivity and social inhibition | Up to six weeks and six months after randomization
  Changes in type d personality and its traits negative affectivity and social inhibition assessed by the Distressed Scale (DS)-14 within and between the two treatment arms. Scores range 0-28, higher scores indicate more symptoms
Changes in quality of life | Up to six weeks and six months after randomization
  Changes in quality of life assessed by the Short Form (SF) 12 within and between the two treatment arms. Scores range 1-100, lower scores indicate lower quality of life
Changes in Bergen Insomnia Scale scores | Up to six weeks and six months after randomization
  Changes in Bergen Insomnia Scale scores assessed by the Bergen Insomnia Scale within and between the two treatment arms. Scores range 0-42, higher scores indicate more symptoms
Changes in C-reactive Protein (CRP) | Up to six weeks and six months after randomization
  Changes in C-reactive Protein (CRP) measured in blood within and between the two treatment arms. Values range 0 to >20, higher values indicate more subclinical inflammation

CONTACTS AND LOCATIONS:
Locations (2):
- Norway (2):
  - Hospital of Vestfold, Tønsberg, Vestfold and Telemark County
  - Vestre Viken Trust Drammen hospital, Drammen, Viken County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tunheim K, Papageorgiou C, Lie HC, Munkhaugen J, Dammen T. Experiences of the attention training technique delivered in groups as treatment for anxiety and depression in patients with coronary heart disease: a qualitative study. BMC Psychiatry. 2025 Jun 3;25(1):573. doi: 10.1186/s12888-025-07027-4. PMID 40461992
- [Derived] Dammen T, Tunheim K, Munkhaugen J, Klungsoyr O, Papageorgiou C. Attention training technique delivered in groups as treatment for anxiety and depression in patients with coronary heart disease: study protocol for a waiting-list randomized controlled trial. Front Psychol. 2023 Sep 18;14:1226539. doi: 10.3389/fpsyg.2023.1226539. eCollection 2023. PMID 37790218